# EFFECTIVENESS OF SCREENING AND BRIEF INTERVENTIONS FOR ALCOHOL AND TOBACCO DURING BREAST CANCER TREATMENT

NCT03371732

15/10/2015

#### PROTOCOL SUMMARY

## Scientific background

It is now well-documented that alcohol and tobacco reduce the effectiveness of treatments, increase their side effects, seem to promote recurring and/or secondary cancers and have effects on the quality of life of patients treated for a cancer pathology. Breast cancer is a common disease for which more than 80% of patients will still be in remission 5 years after the disease. These women constitute a population which can greatly benefit from assistance concerning the adoption of beneficial behaviours for health or from assistance in reducing behavioural risks, particularly related to alcohol and tobacco. The 2014-2019 Cancer Plan emphasises the need to facilitate access to care for patients with problematic substance use. A programme of early intervention practices (spotting, detection, brief intervention and referral) focusing specifically on the oncological context can therefore be a public health approach aimed at reducing the harmful consequences of substance misuse and at improving the prognosis and quality of life of at-risk consumers.

## **Primary objectives**

- Evaluate the effects of the implementation in clinical routine of a programme of identification, detection, and brief interventions with women treated for breast cancer, with high-risk consumption behaviours (alcohol and tobacco) and evaluate the effects of device implantation
- Evaluate the effectiveness of a brief motivational intervention in the short and medium term compared to a basic standard counselling type intervention;

### **Procedure**

Prospective randomised pilot study with control group. Inclusion of 200 patients followed for a first breast cancer and having a positive AUDIT-C score and/or tobacco consumption.

- At the time of the medical consultation, the patient will be offered the possibility of being contacted for screening for psychological distress and her lifestyle concerning alcohol and tobacco, by a trained psychology research assistant. The patient will also give her consent to complete an assessment which will take place before the caregiver interview.
- A certain number of psychological and behavioural variables will be informed via an online questionnaire: screening for alcohol and tobacco consumption, diagnoses of substance-related disorders, anxiety-depressive disorders, quality of life, emotional distress, consumption of patient's family and close friends, self-efficacy and perceived importance, empowerment, and motivation to change will be taken into account. Socio-demographic,

medical and past interventions related to problematic PAS consumption will also be provided.

- Interview conducted by a psychology research assistant trained in the detection of distress, the identification of high-risk behaviour and in brief intervention. Review of the psychoactive substance (PAS) consumption detection results and brief motivational intervention (G1) or educational advice on alcohol and tobacco (G2).

Three months and 6 months (T4) after the brief intervention, the quantitative evaluation of all the psychological and medical variables (except for aspect 1 disorders and socio-demographic data) will be repeated.

# **Anticipated results**

#### Demonstration of:

- the effectiveness of brief motivational-type intervention strategies on high-risk consumption behaviours in patients treated for breast cancer; psychosocial risk factors involved in the maintenance of problematic consumption or in the rapid resumption of consumption behaviours.

The advantage of implementing this type of procedure is on the one hand to be able to set up an early system of access to care, in particular by promoting the care of the most vulnerable groups. It also aims to promote the systematic screening of all psycho-social needs, including an exploration of the patient's lifestyle. This approach is intended to develop a culture of prevention and risk reduction during the care of women treated for breast cancer. Moreover, this type of programme can drive a change in the representations of caregivers in oncology concerning addictive behaviour. Specific training modules can then be offered.